CLINICAL TRIAL: NCT00868933
Title: Low Glycemic Index Dietary Intervention Program in Nonalcoholic Fatty Liver Disease - A Randomized Controlled Trial
Brief Title: Low Glycemic Index Dietary Intervention Program in Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Henry LY Chan, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NAFLD-Diet
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

ARMS (2):
- Low glycemic index dietary intervention program (Active Comparator): The intervention group involves dietary advice and monitoring. No drug or invasive procedure is involved.
  Interventions: Other: Low glycemic index dietary intervention program
- Simple lifestyle advice (Placebo Comparator): The control group receives lifestyle advice from a clinician, and the clinical care is not inferior to current practice.
  Interventions: Other: simple lifestyle advice

INTERVENTIONS:
Other: Low glycemic index dietary intervention program — The intervention group involves dietary advice and monitoring. No drug or invasive procedure is involved.
  Arms: Low glycemic index dietary intervention program
Other: simple lifestyle advice — The control group receives lifestyle advice from a clinician, and the clinical care is not inferior to current practice.
  Arms: Simple lifestyle advice

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is the most common chronic liver disease in affluent countries. It may progress to cirrhosis and liver cancer. At present, there is no approved drug for NAFLD. Although healthy diet and exercise is often recommended, there is little supportive evidence. Therefore, the investigators plan to conduct a randomized controlled trial comparing a low glycemic index dietary intervention program and simple lifestyle advice in NAFLD patients. The primary endpoint is resolution of NAFLD. Non-invasive tests will be used to assess the study subjects. Proton-magnetic resonance spectroscopy is used to quantify hepatic triglyceride content, and transient elastography is used to quantify liver fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Fatty liver by proton-magnetic resonance spectroscopy, defined as hepatic triglyceride content 5% or above
* Serum alanine aminotransferase (ALT) above 30 U/L in men and 19 U/L in women
* Informed written consent obtained

Exclusion Criteria:

* Positive hepatitis B surface antigen, anti-hepatitis C virus antibody, or anti-nuclear antibody titer above 1/160
* Alcohol consumption above 30 g per week in men or 20 g per week in women
* Alanine aminotransferase (ALT) above 10 times the upper limit of normal
* Liver decompensation, as evidenced by bilirubin above 50 µmol/l, platelet count below 100 × 10e9/l, prothrombin time above 1.3 times the upper limit of normal, albumin below 35 g/l, presence of ascites or varices
* Evidence of hepatocellular carcinoma
* Terminal illness or cancer, unless in complete remission for more than 5 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2009-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Resolution of NAFLD by proton-magnetic resonance spectroscopy | Month 12

SECONDARY OUTCOMES:
Partial resolution of NAFLD | Month 12
Visceral fat measurement | Month 12
Liver fibrosis by transient elastography | Month 12
Metabolic endpoints | Month 12

CONTACTS AND LOCATIONS:
Locations (1):
- Cheng Suen Man Shook Hepatitis Center, Institute of Digestive Disease, The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong SAR, China

REFERENCES:
- [Background] Farrell GC, Larter CZ. Nonalcoholic fatty liver disease: from steatosis to cirrhosis. Hepatology. 2006 Feb;43(2 Suppl 1):S99-S112. doi: 10.1002/hep.20973. PMID 16447287
- [Background] Wong VW, Chan HL, Hui AY, Chan KF, Liew CT, Chan FK, Sung JJ. Clinical and histological features of non-alcoholic fatty liver disease in Hong Kong Chinese. Aliment Pharmacol Ther. 2004 Jul 1;20(1):45-9. doi: 10.1111/j.1365-2036.2004.02012.x. PMID 15225170
- [Background] Wong VW, Wong GL, Chim AM, Tse AM, Tsang SW, Hui AY, Choi PC, Chan AW, So WY, Chan FK, Sung JJ, Chan HL. Validation of the NAFLD fibrosis score in a Chinese population with low prevalence of advanced fibrosis. Am J Gastroenterol. 2008 Jul;103(7):1682-8. doi: 10.1111/j.1572-0241.2008.01933.x. Epub 2008 Jul 4. PMID 18616651
- [Background] Hui AY, Wong VW, Chan HL, Liew CT, Chan JL, Chan FK, Sung JJ. Histological progression of non-alcoholic fatty liver disease in Chinese patients. Aliment Pharmacol Ther. 2005 Feb 15;21(4):407-13. doi: 10.1111/j.1365-2036.2005.02334.x. PMID 15709991
- [Background] Caldwell SH, Oelsner DH, Iezzoni JC, Hespenheide EE, Battle EH, Driscoll CJ. Cryptogenic cirrhosis: clinical characterization and risk factors for underlying disease. Hepatology. 1999 Mar;29(3):664-9. doi: 10.1002/hep.510290347. PMID 10051466
- [Background] Wong VW, Hui AY, Tsang SW, Chan JL, Tse AM, Chan KF, So WY, Cheng AY, Ng WF, Wong GL, Sung JJ, Chan HL. Metabolic and adipokine profile of Chinese patients with nonalcoholic fatty liver disease. Clin Gastroenterol Hepatol. 2006 Sep;4(9):1154-61. doi: 10.1016/j.cgh.2006.06.011. Epub 2006 Aug 14. PMID 16904946
- [Background] Targher G, Bertolini L, Rodella S, Tessari R, Zenari L, Lippi G, Arcaro G. Nonalcoholic fatty liver disease is independently associated with an increased incidence of cardiovascular events in type 2 diabetic patients. Diabetes Care. 2007 Aug;30(8):2119-21. doi: 10.2337/dc07-0349. Epub 2007 May 22. No abstract available. PMID 17519430
- [Background] Wong VW, Hui AY, Tsang SW, Chan JL, Wong GL, Chan AW, So WY, Cheng AY, Tong PC, Chan FK, Sung JJ, Chan HL. Prevalence of undiagnosed diabetes and postchallenge hyperglycaemia in Chinese patients with non-alcoholic fatty liver disease. Aliment Pharmacol Ther. 2006 Oct 15;24(8):1215-22. doi: 10.1111/j.1365-2036.2006.03112.x. PMID 17014580
- [Background] Belfort R, Harrison SA, Brown K, Darland C, Finch J, Hardies J, Balas B, Gastaldelli A, Tio F, Pulcini J, Berria R, Ma JZ, Dwivedi S, Havranek R, Fincke C, DeFronzo R, Bannayan GA, Schenker S, Cusi K. A placebo-controlled trial of pioglitazone in subjects with nonalcoholic steatohepatitis. N Engl J Med. 2006 Nov 30;355(22):2297-307. doi: 10.1056/NEJMoa060326. PMID 17135584
- [Background] Nissen SE, Wolski K. Effect of rosiglitazone on the risk of myocardial infarction and death from cardiovascular causes. N Engl J Med. 2007 Jun 14;356(24):2457-71. doi: 10.1056/NEJMoa072761. Epub 2007 May 21. PMID 17517853
- [Background] Chan HL, de Silva HJ, Leung NW, Lim SG, Farrell GC; Asia-Pacific Working Party on NAFLD. How should we manage patients with non-alcoholic fatty liver disease in 2007? J Gastroenterol Hepatol. 2007 Jun;22(6):801-8. doi: 10.1111/j.1440-1746.2007.04977.x. PMID 17565632
- [Background] Chan HL, Wong VW. Can dietetic intervention for obesity ever succeed in real life? J Gastroenterol Hepatol. 2007 Apr;22(4):459-60. doi: 10.1111/j.1440-1746.2007.04931.x. No abstract available. PMID 17376032
- [Background] Ludwig DS. Clinical update: the low-glycaemic-index diet. Lancet. 2007 Mar 17;369(9565):890-2. doi: 10.1016/S0140-6736(07)60427-9. No abstract available. PMID 17368136
- [Background] Woo J, Sea MM, Tong P, Ko GT, Lee Z, Chan J, Chow FC. Effectiveness of a lifestyle modification programme in weight maintenance in obese subjects after cessation of treatment with Orlistat. J Eval Clin Pract. 2007 Dec;13(6):853-9. doi: 10.1111/j.1365-2753.2006.00758.x. PMID 18070255
- [Derived] Shen J, Wong GL, Chan HL, Chan RS, Chan HY, Chu WC, Cheung BH, Yeung DK, Li LS, Sea MM, Woo J, Wong VW. PNPLA3 gene polymorphism and response to lifestyle modification in patients with nonalcoholic fatty liver disease. J Gastroenterol Hepatol. 2015 Jan;30(1):139-46. doi: 10.1111/jgh.12656. PMID 25040896
- [Derived] Wong VW, Chan RS, Wong GL, Cheung BH, Chu WC, Yeung DK, Chim AM, Lai JW, Li LS, Sea MM, Chan FK, Sung JJ, Woo J, Chan HL. Community-based lifestyle modification programme for non-alcoholic fatty liver disease: a randomized controlled trial. J Hepatol. 2013 Sep;59(3):536-42. doi: 10.1016/j.jhep.2013.04.013. Epub 2013 Apr 23. PMID 23623998